CLINICAL TRIAL: NCT07000266
Title: Recovering Coronary Microvascular Obstruction With Supersaturated Oxygen Therapy in ST-segment Elevation Myocardial Infarction (STEMI) Patients: The RECOVERY Study
Brief Title: The RECOVERY Study: Using Supersaturated Oxygen Therapy To Treat Small Vessel Blockages After a Heart Attack
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacio Privada Mon Clinic Barcelona (Other)
Collaborators: Zoll Medical Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-ZOL-501
Record Dates: First submitted 2025-05-08; First posted 2025-06-02 (Actual); Last update posted 2025-06-02 (Actual); Status verified 2025-05

CONDITIONS: Anterior STEMI
Keywords: TherOx DownStream System; Microvascular obstruction; Supersaturated oxygen therapy; SSO2; Percutaneous Coronary Intervention (PCI)
MeSH Terms: interventions — Percutaneous Coronary Intervention; Diagnostic Imaging

STUDY DESIGN:
Intervention Model Description: This is an investigator-initiated, post-market clinical investigation, interventional, prospective, randomized, controlled, open-label, monocenter study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Percutaneous Coronary Intervention (PCI) plus supersaturated oxygen (SSO2) therapy (Experimental): Treatment group
  Interventions: Procedure: Percutaneous Coronary Intervention (PCI); Diagnostic Test: Diagnostic Imaging; Device: Device Treatment; Procedure: Follow-up at 30 days; Procedure: Follow-up at 60 days; Procedure: Follow-up at 12 months
- Standard Percutaneous Coronary Intervention (PCI) (Experimental): Control group
  Interventions: Procedure: Percutaneous Coronary Intervention (PCI); Diagnostic Test: Diagnostic Imaging; Procedure: Follow-up at 30 days; Procedure: Follow-up at 60 days; Procedure: Follow-up at 12 months

INTERVENTIONS:
Procedure: Percutaneous Coronary Intervention (PCI) — Standard PCI intervention
Diagnostic Test: Diagnostic Imaging — Cardiac Magnetic Ressonance (CMR) and hospital discharge
Device: Device Treatment — SSO2 therapy
  Arms: Standard Percutaneous Coronary Intervention (PCI) plus supersaturated oxygen (SSO2) therapy
Procedure: Follow-up at 30 days — Remote (phone) follow-up at 30 days
Procedure: Follow-up at 60 days — In person follow-up at 60 days
Procedure: Follow-up at 12 months — Remote (phone) follow-up at 12 months

SUMMARY:
The study tests whether adding supersaturated oxygen (SSO₂) therapy to standard stent treatment can improve heart recovery after a major heart attack (anterior STEMI). Adults treated within 6 hours of symptoms will be randomly assigned to receive either standard care or standard care plus SSO₂. The goal is to see if SSO₂ reduces damage to small heart vessels. Heart function will be checked immediately, after one hour, and again at six months. Follow-up visits will track recovery for up to a year.

DETAILED DESCRIPTION:
This is an investigator-initiated, post-market clinical investigation, interventional, prospective, randomized, controlled, open-label, monocenter study, in subjects with anterior STEMI with two parallel arms comparing the efficacy of SSO2 with standard PCI and standard PCI alone on reduction of microvascular resistances (Rµ)

Patients will be ≥ 18 years old and diagnosed with a first anterior STEMI requiring stent placement, symptoms duration of ≤ 6 hours and culprit lesion in the left anterior descending (LAD) artery with a TIMI (Thrombolysis In Myocardial Infarction) flow 0 or 1 without collateral circulation.

Patients who provide informed consent will be treated with primary PCI with stenting. Once the coronary blood flow is re-established, and after general and angiographic inclusion and exclusion criteria are confirmed, patients will be randomized and enrolled in the study.

A total number of 20 patients will be randomized (1:1) to SSO2 plus PCI arm or standard PCI control arm. Once randomized, SSO2 arm patients will receive SSO2 therapy inside the catheterization laboratory, meanwhile patients randomized in the standard arm will not receive further treatment beyond standard of care.

For both arms, coronary invasive measurements will be performed immediately and 60 minutes after coronary blood flow restoration and then at 6 months timepoint. Baseline clinical and procedural variables will be collected. There will be a clinical follow-up at 30 days ± 7 days, 6 months ± 1 month and 1 year ± 1 month after index event.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be ≥ 18 years of age
2. Anterior STEMI (ECG with persistent elevation ≥ 2 mm (0.2 mV) in 2 or more contiguous anterior precordial leads (V2, V3, V4) in men or ≥ 1.5 mm (0.15 mV) in women.
3. Symptoms consistent with myocardial ischemia (persistent chest pain, dyspnea, nauseas/vomiting, fatigue, palpitations or syncope) present for ≤ 6 hours.
4. Provision of informed consent by patient
5. Culprit lesion in proximal or mid LAD.
6. Pre-PCI TIMI flow 0-1.
7. The patient is eligible for primary PCI.
8. Successful PCI of a proximal or mid LAD lesion with commercially available coronary stents and achievement of TIMI 2 or 3 flow
9. Expected ability to place the catheter in the left main coronary ostium to deliver SSO2 therapy with stable and coaxial alignment.

Exclusion Criteria:

1. Previous MI, PCI or CABG occurred before index procedure.
2. Previous history of stroke, transient ischemic attack (TIA) or reversible ischemic neurological deficit within last 6 months.
3. Known severe kidney disease (eGFR <=30 mL/min/1.73) and/or hemodialysis.
4. Known coagulopathy.
5. Known ongoing anticoagulant treatment.
6. Known large pericardial effusion or cardiac tamponade.
7. Known allergies to polyurethanes, PET or stainless steel.
8. Unconscious at presentation.
9. Need for circulatory support.
10. Need for invasive mechanical ventilation.
11. Need for temporal intravenous pacemaker.
12. Cardiopulmonary resuscitation (CPR) cardiac arrest ≥ 5 minutes whom baseline neurologic status is not present.
13. Patients confirmed as pregnant.
14. Active participation in another drug or device investigational trial.
15. Known contraindication for adenosine administration (severe asthma, complicated AV block, critical aortic stenosis, severe cardiac arrhythmias, severe valve diseases).
16. Patient not suitable for femoral access.
17. Patients with mechanical complications of STEMI.
18. Known epicardial stenosis on LAD lesion after stent placement that restricts flow with the SSO2 delivery catheter in place.
19. Ipsilateral insertion of a second sheath in a single femoral artery for SuperSaturated Oxygen Therapy is strictly contraindicated
20. Presence of an intra-aortic balloon pump.
21. Presence of a post-intervention non-stented coronary dissection or perforation.
22. Cardiac valvular stenosis or insufficiency, pericardial disease or non-ischemic cardiomyopathy.
23. Cardiogenic shock.
24. Subjects with ventricular pseudoaneurysm, VSD, or severe mitral valve regurgitation (with or without papillary muscle rupture).
25. Hemoglobin < 10 g/dL.
26. Gastrointestinal or genitourinary bleeding within the last two months, or any major surgery (including CABG) within six weeks of procedure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-23 (Actual); Primary Completion 2027-05-16 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Effect of SSO2 on microvascular resistances (Rµ) | 60 minutes after primary PCI
  Superiority in % of patients without microvascular dysfunction (defined as microvascular resistance >500 WU) of SSO2 arm versus standard of care (90% of patients with microvascular dysfunction in the control arm vs. 30% in the SSO2 arm)

SECONDARY OUTCOMES:
Effect of SSO2 on absolute coronary flow (Q) | At 60 minutes and at 6 months after primary PCI
  Absolute coronary flow (Q): difference in Q, between the SSO2 arm and the standard PCI control arm, evaluated with invasive coronary measurement.
Effect of SSO2 on the index of microvascular resistance (IMR) | Within 5 minutes after primary PCI, at 60 minutes after primary PCI and at 6 months after primary PCI
  Microvascular resistances (Rµ): difference in (Rµ) between the SSO2 arm and the standard PCI control arm, evaluated with invasive coronary measurement.
Effect of SSO2 on the index of microvascular resistance (IMR) | Within 5 minutes after primary PCI, at 60 minutes after primary PCI and at 6 months after primary PCI
  Index of microvascular resistance (IMR): difference in IMR between the SSO2 arm and the standard PCI control arm, evaluated with invasive coronary measurement.
Effect of SSO2 on the coronary flow reserve (CFR) | Within 5 minutes after primary PCI, at 60 minutes after PCI and at 6 months after primary PCI
  Coronary flow reserve (CFR): difference in CFR between the SSO2 arm and the standard PCI control arm, evaluated with invasive coronary measurement.
Effect of SSO2 on the microvascular resistance reserve (MRR) | Within 5 minutes after primary PCI, at 60 minutes after primary PCI and at 6 months after primary PCI
  Microvascular resistance reserve (MRR): difference in MRR between the SSO2 arm and the standard PCI control arm, evaluated with invasive coronary measurement.
Effect of SSO2 on infarct size and microvascular obstruction at CMR | At CMR 3-5 days after primary PCI
  Quantification of infarct size as a percentage of left ventricular mass using late gadolinium enhancement (LGE) and assessment of microvascular obstruction (MVO) presence and extent.
Risk of predefined major cardiovascular adverse events (MACE) during treatment and follow-up | During treatment, during follow-up at 30 days, 60 days and 12 months follow-ups
  Time from randomization to the first occurrence of any event in the predefined MACE composite per patient.
Risk of predefined major cardiovascular adverse events (MACE) during treatment and follow-up | At at 30 days, 6 months and 1 year follow-ups after index PCI
  Per-patient rate of composite MACE events (first and subsequent)

OTHER OUTCOMES:
Effect of SSO2 on ventricular remodeling | From baseline to follow-up CMR
  Proportion of patients with adverse ventricular remodeling, defined as a Δ ≥20% in end-diastolic volume (EDV) or a Δ ≥15% in end-systolic volume (ESV), with additional assessment of myocardial tissue characteristics using T2-weighted imaging and LGE.
Effect of SSO2 on left ventricular hypertrophy | At CMR 3-5 days after primary PCI
  Proportion of patients with left ventricular hypertrophy in the SSO2 therapy arm compared to the standard PCI control arm, as assessed by CMR. Left ventricular hypertrophy is considered for masses above 106.2 g/m2 for men and 84.6 g/m2 in women

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No